CLINICAL TRIAL: NCT03439228
Title: To Brace or Not to Brace for Single Level Lumbar Fusion: a Pilot Prospective Randomized Controlled Trial
Brief Title: To Brace or Not to Brace for Single Level Lumbar Fusion Pilot
Acronym: BRACE Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); DJO Incorporated (Industry); Stryker Canada LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3478
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Spondylosis; Fusion of Spine
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brace (Experimental): Lumbar brace wear prescribed for 3 months post-operation
  Interventions: Device: Lumbar brace
- No brace (No Intervention): No lumbar brace prescribed

INTERVENTIONS:
Device: Lumbar brace — 3 months of lumbar brace wear
  Arms: Brace

SUMMARY:
The use of a lumbar brace following single-level lumbar fusion for degenerative spondylosis (non-traumatic) is variable between surgeons. Some surgeons prefer to prescribe a brace and others do not. There is a lack of guidelines and evidence to support either treatment option. The purpose of this study is to assess feasibility and collect preliminary data to conduct a larger, definitive trial to provide evidence as to whether prescribing a brace or not results in better or equal outcomes. Imaging by CT scan, one year after surgery, will be used to analyze bone fusion (healing), and functional and pain scores from patients during their recovery will be compared to identify differences between patients who wore a brace and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Single-level lumbar instrumented postero-lateral fusion from L2-L5
* Life expectancy greater than 2 years

Exclusion Criteria:

* Previous lumbar surgery
* Spine tumour/cancer
* Documented osteoporosis
* High grade (3 or 4) spondylolisthesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of enrolment | 12 months
  Feasibility measure to assess pilot project design. Assess ability to recruit 2 patients per month.
Rate of study completion | 12 months
  Feasibility measure to assess pilot project design. Evaluate study visit and study completion rates.

SECONDARY OUTCOMES:
Lumbar bone fusion | 12 months
  Status of bone fusion assessed radiologically by CT scan
Functional Status | 3 months, 6 months, 12 months
  The Oswestry Disability Index
Pain Status | 3 months, 6 months, 12 months
  Visual analog scale (0, no pain to 10, worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksa Cenic, MSc, MD, FRCSC, Principal Investigator — Hamilton Health Sciences and McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No